CLINICAL TRIAL: NCT02578017
Title: ENHANCE Study (ElectroNic Hydroxyurea AdhereNCE): A Strategy to Improve Hydroxyurea Adherence in Patients With Sickle Cell Disease
Brief Title: ElectroNic Hydroxyurea AdhereNCE: A Strategy to Improve Hydroxyurea Adherence in Patients With Sickle Cell Disease
Acronym: ENHANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Susan Creary, Assistant Professor of Pediatric Hematology/Oncology, Nationwide Children's Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NCH14-00163
Record Dates: First submitted 2015-09-23; First posted 2015-10-16 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Hydroxyurea; Adherence
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mobile DOT (Experimental): All Participants will utilize Mobile DOT for 6 months. The Mobile DOT intervention includes: reminder alerts, participant videos, research staff feedback on adherence, and contingency management.
  Interventions: Behavioral: Mobile DOT
- Post-intervention observation (No Intervention): All participants will not receive any additional adherenece intervention after completing the Mobile DOT arm. Participants will be observed for 6 months.

INTERVENTIONS:
Behavioral: Mobile DOT — Mobile DOT is a multi-dimensional tool that uses automated reminders, adherence feedback messages, incentives, and video observation of medication administration.
  Arms: Mobile DOT

SUMMARY:
HU is an FDA approved medication for the treatment of SCD. Many studies have shown that HU can reduce SCD related symptoms, but only 50% of patients take it as often as they should. This limits how much HU can help reduce SCD symptoms.

Researchers are interested to see if electronic directly observed therapy (Mobile DOT), a program that uses cell phone reminder messages, videos, feedback messages, and incentives will help patients with SCD take HU as prescribed.

DETAILED DESCRIPTION:
This is a 12-month, single-arm, cross-over study for pediatric and adolescent patients with SCD who are prescribed HU at Nationwide Children's Hospital in order to compare HU adherence prior to the study, during Mobile Dot use and after using Mobile DOT.

Hydroxyurea (HU) is the only disease-modifying medication for patients with sickle cell disease (SCD). Multiple clinical trials show that HU can reduce SCD-related complications but only 50% of pediatric patients adhere to HU at the rates achieved in clinical trials. This poor adherence limits its clinical effectiveness and results in increased costs and in lower patient-reported quality of life.

An innovative, practical, inexpensive, and efficient strategy is needed to improve HU adherence in pediatric patients with SCD. Electronic directly observed therapy (Mobile DOT) is a pilot-tested, multi-dimensional tool that is a feasible and acceptable strategy and can achieve >90% HU adherence rates in a small cohort of pediatric patients with SCD. This study will provide further testing to confirm if Mobile DOT can improve adherence and improve clinical outcomes in patients with SCD.

Mobile DOT uses patients' smart phones and computers to provide electronic reminder alerts and to video-record patients' daily HU administrations. Patients are provided with text (SMS) messages, e-mails, and phone call communications to encourage adherence and they receive monetary incentives when they reach adherence goals.

Researchers will determine if video adherence correlates with self-report, biomarker, and refill adherence. Also, surveys will be completed by participants to determine if their self-management skills improve with Mobile DOT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Sickle Cell Disease (SCD), any genotype
* Prescribed HU for at least the previous 6 months
* Plans to receive SCD-related care at Nationwide Children's Hospital for the study duration
* For participants ≥18 years: participant must have access to a smart-phone or computer capable of recording and submitting videos to Mobile DOT
* For participants <18 years: consenting adult must have access to a smart-phone or computer capable of recording and submitting videos to Mobile DOT AND agrees to enter into a mutual agreement to participate in the daily medication administration routine
* Patient and/or consenting adult must speak English
* Access to a working phone (smart phone or landline)

Exclusion Criteria:

* Current chronic transfusion therapy or apheresis

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2014-07; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Achievement of ≥80% HU adherence | 12 months
  Compare the number of participants who achieve ≥80% HU adherence when patients receive Mobile DOT to the 6 months prior to study entry.

SECONDARY OUTCOMES:
Correlation of video observation adherence with other measures of adherence. | 12 months
  Determine if video observation adherence correlations with biomarker adherence (MCV, HbF, and urine assay), self-report, and refill estimated adherence.
Changes in self-managment skills | 12 months
  To explore adolescent and young adults' self-managment skills using the transition readiness questionnaire before and after mobile DOT.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Creary, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Creary S, Chisolm D, Stanek J, Neville K, Garg U, Hankins JS, O'Brien SH. Measuring hydroxyurea adherence by pharmacy and laboratory data compared with video observation in children with sickle cell disease. Pediatr Blood Cancer. 2020 Aug;67(8):e28250. doi: 10.1002/pbc.28250. Epub 2020 May 9. PMID 32386106
- [Derived] Creary S, Chisolm D, Stanek J, Hankins J, O'Brien SH. A Multidimensional Electronic Hydroxyurea Adherence Intervention for Children With Sickle Cell Disease: Single-Arm Before-After Study. JMIR Mhealth Uhealth. 2019 Aug 8;7(8):e13452. doi: 10.2196/13452. PMID 31397291